CLINICAL TRIAL: NCT05111613
Title: The PEERLESS Study
Acronym: PEERLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inari Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-002
Record Dates: First submitted 2021-10-15; First posted 2021-11-08 (Actual); Results first posted 2025-11-13 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Embolism; Pulmonary Thromboembolism
Keywords: PE; pulmonary embolism; thrombectomy; FlowTriever; CDT; Catheter-Directed Thrombolysis
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Randomized Controlled Trial Cohort - FlowTriever Arm (Active Comparator): Mechanical thrombectomy for pulmonary embolism using the FlowTriever System.
  Interventions: Device: FlowTriever System
- Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm (Active Comparator): Catheter-Directed Thrombolysis for pulmonary embolism (any commercially available CDT system)
  Interventions: Device: Catheter-Directed Thrombolysis
- Non-Randomized Absolute Contraindication to Thrombolytics Cohort (Other): Mechanical thrombectomy for pulmonary embolism using the FlowTriever System.
  Interventions: Device: FlowTriever System

INTERVENTIONS:
Device: Catheter-Directed Thrombolysis — Catheter-Directed Thrombolysis for pulmonary embolism (any commercially available CDT system)
  Arms: Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm
Device: FlowTriever System — Mechanical thrombectomy for pulmonary embolism
  Arms: Non-Randomized Absolute Contraindication to Thrombolytics Cohort; Randomized Controlled Trial Cohort - FlowTriever Arm

SUMMARY:
A prospective, multicenter, randomized controlled trial of the FlowTriever System compared to Catheter-Directed Thrombolysis (CDT) for use in the treatment of acute pulmonary embolism. The trial includes a non-randomized cohort of subjects with an absolute contraindication to thrombolysis.

ELIGIBILITY:
Inclusion Criteria

Subjects must meet each of the following criteria to be included in the study:

* Age ≥ 18 years
* Echo, computed tomographic pulmonary angiography (CTPA), or pulmonary angiographic evidence of any proximal filling defect in at least one main or lobar pulmonary artery
* Including ALL of the following: Clinical signs and symptoms consistent with acute PE, or PESI class III-V, or sPESI ≥1; AND Hemodynamically stable AND; RV dysfunction on echocardiography or CT; AND Any one or more of the following present at the time of diagnosis: Elevated cardiac troponin levels; History of heart failure; History of chronic lung disease; Heart rate ≥110 beats per minute; SBP <100mmHg; Respiratory rate ≥30 breaths per minute; O2 saturation <90%; Syncope related to PE; Elevated Lactate
* Intervention planned to begin within 72 hours of the later of either: confirmed PE diagnosis; OR if transferring from another hospital, arrival at the treating hospital
* Symptom onset within 14 days of confirmed PE diagnosis

Exclusion Criteria

Subjects will be excluded from the study for any of the following criteria:

* Unable to anticoagulate with heparin, enoxaparin or other parenteral antithrombin
* Index presentation with hemodynamic instability that are part of the high-risk PE definition in the ESC Guidelines 2019, including ANY of the following: cardiac arrest; OR systolic BP < 90 mmHg or vasopressors required to achieve a BP ≥90 mmHg despite adequate filling status, AND end-organ hypoperfusion; OR systolic BP < 90 mmHg or systolic BP drop ≥40 mmHg, lasting longer than 15 min and not caused by new-onset arrhythmia, hypovolemia, or sepsis
* Known sensitivity to radiographic contrast agents that, in the Investigator's opinion, cannot be adequately pre-treated
* Imaging evidence or other evidence that suggests, in the opinion of the Investigator, the patient is not appropriate for catheter-based intervention (e.g. inability to navigate to target location, clot limited to segmental/subsegmental distribution, predominately chronic clot)
* Patient has right heart clot in transit identified at baseline screening
* Life expectancy < 30 days (e.g. stage 4 cancer or severe COVID-19 infection), as determined by the Investigator
* Current participation in another drug or device study that, in the Investigator's opinion, would interfere with participation in this study
* Current or history of chronic thromboembolic pulmonary hypertension (CTEPH) or chronic thromboembolic disease (CTED) diagnosis, per ESC 2019 guidelines
* Invasive systolic PA pressure ≥70 mmHg prior to study device entering the body
* Administration of bolus or drip/infusion thrombolytic therapy or mechanical thrombectomy for the index PE event within 48 hours prior to enrollment
* Ventricular arrhythmias refractory to treatment at the time of enrollment
* Known to have heparin-induced thrombocytopenia (HIT)
* Subject has any condition for which, in the opinion of the Investigator, participation would not be in the best interest of the subject (e.g., compromise the well-being or that could prevent, limit, or confound the protocol-specified assessments). This includes a contraindication to use of FlowTriever or CDT System (for example, EKOS System) per local approved labeling
* Subject has previously completed or withdrawn from this study
* Patient unwilling or unable to conduct the follow up visits per protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 692 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wissam Jaber, MD, Principal Investigator — Emory University; Carin Gonsalves, MD, Principal Investigator — Thomas Jefferson University; Stefan Stortecky, MD, Principal Investigator — Bern University Hospital
Locations (60):
- United States (56):
  - Loma Linda University Health, Loma Linda, California
  - Providence St. Joseph Orange, Orange, California
  - Huntington Hospital, Pasadena, California
  - University of Colorado Hospital, Aurora, Colorado
  - Radiology and Imaging Associates, Lakeland, Florida
  - Baptist Health South Florida, Miami, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Tallahassee Memorial Hospital, Tallahassee, Florida
  - University of South Florida Tampa General Hospital, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Ascension Alexian Brothers Medical Center, Elk Grove Village, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Ascension St. Vincent Hospital - Indianapolis, Indianapolis, Indiana
  - Norton Healthcare, Louisville, Kentucky
  - Brigham and Womens Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Ascension St. John Hospital, Detroit, Michigan
  - CentraCare St. Cloud Hospital, Saint Cloud, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Saint Louis University, St Louis, Missouri
  - Virtua Lourdes, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Northwell Health, Bay Shore, New York
  - Gates Vascular Institute, Buffalo, New York
  - NewYork-Presbyterian Columbia University Irving Medical Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina Health, Chapel Hill, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Summa Akron City Hospital, Akron, Ohio
  - Mercy Health West, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - OhioHealth Riverside Methodist Hospital, Columbus, Ohio
  - St. Luke's University Hospital, Bethlehem, Pennsylvania
  - AHN Saint Vincent Hospital, Erie, Pennsylvania
  - UPMC Harrisburg, Harrisburg, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - MUSC Health University Medical Center, Charleston, South Carolina
  - Spartanburg Regional Healthcare System, Spartanburg, South Carolina
  - Lexington Medical Center, West Columbia, South Carolina
  - HCA TriStar Centennial Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas Hospital, Nashville, Tennessee
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - HCA Medical City Heart and Spine, Dallas, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Medical Center, Houston, Texas
  - Methodist Main Hospital, San Antonio, Texas
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Providence Sacred Heart Medical Center, Spokane, Washington
  - Ascension St. Elizabeth Hospital, Appleton, Wisconsin
  - Gundersen Health System, La Crosse, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin
- Germany (3):
  - Universtitaetsklinikum Dusseldorf, Düsseldorf
  - Herzzentrum Leipzig, Leipzig
  - Marien Hospital Wesel GmbH, Wesel
- Inselspital - Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonsalves CF, Gibson CM, Stortecky S, Alvarez RA, Beam DM, Horowitz JM, Silver MJ, Toma C, Rundback JH, Rosenberg SP, Markovitz CD, Tu T, Jaber WA. Randomized controlled trial of mechanical thrombectomy vs catheter-directed thrombolysis for acute hemodynamically stable pulmonary embolism: Rationale and design of the PEERLESS study. Am Heart J. 2023 Dec;266:128-137. doi: 10.1016/j.ahj.2023.09.002. Epub 2023 Sep 12. PMID 37703948
- [Result] Jaber WA, Gonsalves CF, Stortecky S, Horr S, Pappas O, Gandhi RT, Pereira K, Giri J, Khandhar SJ, Ammar KA, Lasorda DM, Stegman B, Busch L, Dexter DJ 2nd, Azene EM, Daga N, Elmasri F, Kunavarapu CR, Rea ME, Rossi JS, Campbell J, Lindquist J, Raskin A, Smith JC, Tamlyn TM, Hernandez GA, Rali P, Schmidt TR, Bruckel JT, Camacho JC, Li J, Selim S, Toma C, Basra SS, Bergmark BA, Khalsa B, Zlotnick DM, Castle J, O'Connor DJ, Gibson CM; PEERLESS Committees and Investigators*. Large-Bore Mechanical Thrombectomy Versus Catheter-Directed Thrombolysis in the Management of Intermediate-Risk Pulmonary Embolism: Primary Results of the PEERLESS Randomized Controlled Trial. Circulation. 2025 Feb 4;151(5):260-273. doi: 10.1161/CIRCULATIONAHA.124.072364. Epub 2024 Oct 29. PMID 39470698

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-Randomized Contraindication to Thrombolytics Cohort: Mechanical thrombectomy for pulmonary embolism using the FlowTriever System.
Period: Overall Study
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Contraindication to Thrombolytics Cohort
Started (Enrolled) | 274 | 276 | 142
Completed | 261 | 255 | 126
Not Completed | 13 | 21 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort | Total
Number analyzed (Participants) | 274 | 276 | 142 | 692
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.7 (13.0) | 61.2 (14.8) | 64.3 (13.9) | 62.8 (14.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125 | 134 | 64 | 323
  Male | 149 | 142 | 78 | 369
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 184 | 193 | 91 | 468
  Black or African American | 67 | 56 | 24 | 147
  Other/multiple | 3 | 7 | 4 | 14
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 3 | 1 | 4
  Unavailable | 20 | 17 | 20 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Subject reported ethnicity was unavailable in 25 subjects in the Randomized Controlled Trial Cohort - FlowTriever Arm, 26 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm, and 20 subjects in the non-randomized cohort.
  Participants
    Hispanic or Latino: number analyzed (Participants) | 249 | 250 | 122 | 621
    Hispanic or Latino | 13 | 27 | 21 | 61
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Data missing for one subject in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm and one subject in the non-randomized cohort.
  kg/m^2
    number analyzed (Participants) | 274 | 275 | 141 | 690
    (all) | 34.5 (8.6) | 36.3 (9.4) | 32.0 (6.7) | 34.7 (8.7)
History of cancer [Count of Participants; unit: Participants] | 56 | 56 | 51 | 163
Active cancer [Count of Participants; unit: Participants] | 13 | 17 | 39 | 69
Prior pulmonary embolism [Count of Participants; unit: Participants] | 41 | 31 | 12 | 84
History of pulmonary hypertension [Count of Participants; unit: Participants] | 6 | 5 | 7 | 18
Prior deep vein thrombosis [Count of Participants; unit: Participants] | 60 | 58 | 25 | 143
Concomitant deep vein thrombosis [Count of Participants; unit: Participants] | 178 | 168 | 90 | 436
History of bleeding [Count of Participants; unit: Participants] | 5 | 9 | 31 | 45
Active bleeding preprocedure [Count of Participants; unit: Participants] | 0 | 2 | 12 | 14
Anemia [Count of Participants; unit: Participants] | 21 | 27 | 47 | 95
History of renal disease [Count of Participants; unit: Participants] | 28 | 33 | 29 | 90
Renal dysfunction (CrCL 30-60 mL/min) [Count of Participants; unit: Participants] | 43 | 45 | 33 | 121
Recent surgery (within 3 weeks) [Count of Participants; unit: Participants] | 22 | 12 | 48 | 82
Recent trauma (within 3 weeks) [Count of Participants; unit: Participants] | 8 | 7 | 18 | 33
Prior cerebrovascular accident [Count of Participants; unit: Participants] | 7 | 8 | 17 | 32
Relative contraindication to thrombolytics [Count of Participants; unit: Participants] — Categories are not mutually exclusive; 11 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm had a total of 12 relative contraindications. Population: Data for this Baseline Measure were only collected for participants in the Randomized Controlled Trial Cohorts and were not available for participants in the Non-Randomized Absolute Contraindication to Thrombolytics Cohort.
  Participants
    Total: number analyzed (Participants) | 274 | 276 | 0 | 550
    Total | 12 | 11 | 0 | 23
    Anemia (hemoglobin <10 g/dL): number analyzed (Participants) | 274 | 276 | 0 | 550
    Anemia (hemoglobin <10 g/dL) | 3 | 5 | 0 | 8
    Oral anticoagulation, except for aspirin: number analyzed (Participants) | 274 | 276 | 0 | 550
    Oral anticoagulation, except for aspirin | 4 | 3 | 0 | 7
    Therapeutic LMWH within 24 hours: number analyzed (Participants) | 274 | 276 | 0 | 550
    Therapeutic LMWH within 24 hours | 4 | 2 | 0 | 6
    Refractory hypertension (SBP >180 mmHg or DBP >110 mmHg on two confirmed measurements: number analyzed (Participants) | 274 | 276 | 0 | 550
    Refractory hypertension (SBP >180 mmHg or DBP >110 mmHg on two confirmed measurements | 1 | 2 | 0 | 3
Absolute contraindication to thrombolytics [Count of Participants; unit: Participants] — Categories are not mutually exclusive. Population: Data for this Baseline Measure were only collected for participants in the Non-Randomized Absolute Contraindication to Thrombolytics Cohort and were not available for participants in the Randomized Controlled Trial Cohorts.
  Participants
    Total: number analyzed (Participants) | 0 | 0 | 142 | 142
    Total | 0 | 0 | 142 | 142
    Any other condition on the product label for use by local standard and investigator discretion: number analyzed (Participants) | 0 | 0 | 142 | 142
    Any other condition on the product label for use by local standard and investigator discretion | 0 | 0 | 62 | 62
    Recent (3 months) intracranial or intraspinal surgery or serious head trauma: number analyzed (Participants) | 0 | 0 | 142 | 142
    Recent (3 months) intracranial or intraspinal surgery or serious head trauma | 0 | 0 | 32 | 32
    Presence of intracranial conditions such as neoplasms, arteriovenous malformations, or aneurysms: number analyzed (Participants) | 0 | 0 | 142 | 142
    Presence of intracranial conditions such as neoplasms, arteriovenous malformations, or aneurysms | 0 | 0 | 24 | 24
    Active internal bleeding, excluding menses: number analyzed (Participants) | 0 | 0 | 142 | 142
    Active internal bleeding, excluding menses | 0 | 0 | 12 | 12
    History of hemorrhagic stroke or stroke of unknown origin: number analyzed (Participants) | 0 | 0 | 142 | 142
    History of hemorrhagic stroke or stroke of unknown origin | 0 | 0 | 10 | 10
    Bleeding diathesis: number analyzed (Participants) | 0 | 0 | 142 | 142
    Bleeding diathesis | 0 | 0 | 10 | 10
    Severe uncontrolled hypertension: number analyzed (Participants) | 0 | 0 | 142 | 142
    Severe uncontrolled hypertension | 0 | 0 | 5 | 5
    Ischemic stroke in the previous 6 months: number analyzed (Participants) | 0 | 0 | 142 | 142
    Ischemic stroke in the previous 6 months | 0 | 0 | 4 | 4
    Aortic dissection: number analyzed (Participants) | 0 | 0 | 142 | 142
    Aortic dissection | 0 | 0 | 2 | 2
VTE-BLEED score [Mean (Standard Deviation); unit: units on a scale] — The VTE-BLEED score is a clinical tool used to estimate the risk of bleeding in subjects receiving long-term anticoagulation treatment for venous thromboembolism (VTE). It helps clinicians identify individuals who may be at increased risk of bleeding and can aid in making informed decisions about anticoagulation strategies. Scores range from 0 to 9. A low score (typically <2) suggests a lower risk of bleeding, while a higher score indicates a greater risk of bleeding.
  units on a scale | 1.55 (1.30) | 1.56 (1.31) | 2.77 (1.78) | 1.8 (1.49)
VTE-BLEED score [Count of Participants; unit: Participants]
  Score >=2 | 68 | 77 | 81 | 226
  Score <2 | 206 | 199 | 61 | 466
sPESI score [Mean (Standard Deviation); unit: units on a scale] — The simplified Pulmonary Embolism Severity Index (sPESI) score is a tool used to classify the risk of death and complications in subjects with pulmonary embolism (PE). The scale ranges from 0 to 6, with higher values indicating increased risk of death and complications. Population: Data unavailable in 1 subject in the Randomized Controlled Trial Cohort - FlowTriever Arm.
  units on a scale
    number analyzed (Participants) | 273 | 276 | 142 | 691
    (all) | 1.3 (1.1) | 1.3 (1.1) | 1.7 (1.1) | 1.4 (1.1)
sPESI score [Count of Participants; unit: Participants] — Population: Data unavailable in 1 subject in the Randomized Controlled Trial Cohort - FlowTriever Arm.
  Participants
    number analyzed (Participants) | 273 | 276 | 142 | 691
    Score >=1 | 203 | 213 | 128 | 544
    Score =0 | 70 | 63 | 14 | 147
Intermediate risk PE [Count of Participants; unit: Participants] — All enrolled subjects were required by protocol to have intermediate-risk PE per European Society of Cardiology (ESC) guidelines (hemodynamic stability and RV dilatation on imaging), and subjects enrolled before protocol version 3.0 were required to have elevated cardiac troponin levels (intermediate-high-risk PE per ESC criteria).
  Participants
    Intermediate-high-risk PE | 256 | 265 | 128 | 649
    Intermediate-low-risk PE | 18 | 11 | 14 | 43
Duration of symptoms, days [Mean (Standard Deviation); unit: days] | 2.9 (2.8) | 3.5 (3.3) | 2.8 (2.8) | 3.1 (3.0)
Elevated cardiac troponin levels [Count of Participants; unit: Participants] | 256 | 265 | 128 | 649
Most central PE location at screening [Count of Participants; unit: Participants]
  Saddle | 104 | 109 | 58 | 271
  Main pulmonary artery | 143 | 143 | 76 | 362
  Lobar | 27 | 24 | 8 | 59
Right bundle branch block [Count of Participants; unit: Participants] | 39 | 36 | 22 | 97
Heart rate, bpm [Mean (Standard Deviation); unit: beats per minute] | 107.2 (17.1) | 111.6 (20.2) | 108.9 (17.2) | 109.3 (18.5)
Respiratory rate, rpm [Mean (Standard Deviation); unit: respirations per minute] — Population: Data unavailable for 1 subject in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm and 1 subject in the non-randomized cohort.
  respirations per minute
    number analyzed (Participants) | 274 | 275 | 141 | 690
    (all) | 22.2 (6.7) | 22.4 (5.9) | 23.1 (6.7) | 22.5 (6.4)
Systolic blood pressure at diagnosis, mmHg [Mean (Standard Deviation); unit: mmHg] — Population: Data unavailable for 1 subject in the non-randomized cohort.
  mmHg
    number analyzed (Participants) | 274 | 276 | 141 | 691
    (all) | 134.0 (22.4) | 132.1 (21.7) | 127.7 (23.7) | 132.0 (22.5)
Diastolic blood pressure at diagnosis, mmHg [Mean (Standard Deviation); unit: mmHg] — Population: Data unavailable for 1 subject in the non-randomized cohort.
  mmHg
    number analyzed (Participants) | 274 | 276 | 141 | 691
    (all) | 83.8 (14.7) | 84.1 (14.7) | 80.0 (14.6) | 83.2 (14.8)
mMRC dyspnea score [Count of Participants; unit: Participants] — The mMRC scale (modified Medical Research Council) is a subject-reported outcome tool used to assess the impact of breathlessness (dyspnea) on daily activities. It is a self-assessment scale ranging from 0 to 4, where higher scores indicate greater breathlessness. Population: Data unavailable for 3 subjects in the Randomized Controlled Trial Cohort - FlowTriever Arm, 3 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm, and 4 subjects in the non-randomized cohort.
  Participants
    number analyzed (Participants) | 271 | 273 | 138 | 682
    Score 0 - Dyspnea only with strenuous exercise | 16 | 12 | 9 | 37
    Score 1 - Dyspnea when hurrying or walking up a slight hill | 23 | 17 | 5 | 45
    Score 2 - Walks slower than people of same age due to dyspnea or has to stop for breath when walking | 37 | 39 | 13 | 89
    Score 3 - Stops for breath after walking 100 yards (91 m) or after a few minutes | 87 | 79 | 36 | 202
    Score 4 - Too dyspneic to leave house or breathless when dressing | 108 | 126 | 75 | 309
NYHA classification [Count of Participants; unit: Participants] — The NYHA (New York Heart Association) classification is a system that categorizes heart failure symptoms based on severity and physical activity limitations. The scale ranges from I to IV, with higher values denoting worse functional capacity and symptoms. Population: Data unavailable for 2 subjects in the Randomized Controlled Trial Cohort - FlowTriever Arm, 3 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm, and 3 subjects in the non-randomized cohort.
  Participants
    number analyzed (Participants) | 272 | 273 | 139 | 684
    Class I - No limitation of physical activity | 26 | 19 | 13 | 58
    Class II - Slight limitation of physical activity | 54 | 51 | 11 | 116
    Class III - Marked limitation of physical activity | 122 | 127 | 58 | 307
    Class IV - Unable to carry on any physical activity without discomfort | 70 | 76 | 57 | 203
Modified Borg dyspnea score [Mean (Standard Deviation); unit: units on a scale] — The Modified Borg dyspnea score is a tool used to measure and quantify the perceived difficulty of breathing during exercise. It is a numerical scale ranging from 0 (no difficulty) to 10 (maximal difficulty). Population: Data unavailable for 2 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm and 7 subjects in the non-randomized cohort.
  units on a scale
    number analyzed (Participants) | 274 | 274 | 135 | 683
    (all) | 3.12 (2.63) | 3.32 (2.58) | 3.93 (2.96) | 3.36 (2.69)
RV/LV ratio (CTPA or echocardiogram) [Mean (Standard Deviation); unit: ratio] — The RV/LV ratio, or right ventricle to left ventricle ratio, is a measurement of the ratio of the right ventricular diameter to the left ventricular diameter. An elevated RV/LV ratio can suggest that the right ventricle is enlarged, which can be a sign of increased pressure or workload on the right heart, and can be an independent predictor of adverse outcomes, such as mortality, in patients with PE. Population: Data unavailable for 12 subjects in the Randomized Controlled Trial Cohort - FlowTriever Arm, 16 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm, and 14 subjects in the non-randomized cohort.
  ratio
    number analyzed (Participants) | 262 | 260 | 128 | 650
    (all) | 1.27 (0.26) | 1.31 (0.27) | 1.31 (0.33) | 1.29 (0.28)
RV function on echocardiogram [Count of Participants; unit: Participants] — Population: Only subjects with RV function collected at both the Baseline and 24 Hour Visit are reported here, resulting in unavailable data for 96 subjects in the RCT FlowTriever cohort, 105 subjects in the RCT CDT cohort, and 62 subjects in the non-randomized cohort.
  Participants
    number analyzed (Participants) | 178 | 171 | 80 | 429
    Normal | 1 | 0 | 2 | 3
    Mildly reduced | 13 | 11 | 3 | 27
    Moderately reduced | 42 | 41 | 19 | 102
    Severely reduced | 122 | 119 | 56 | 297
Parenteral anticoagulation use at baseline [Count of Participants; unit: Participants]
  UFH and/or LMWH: Total | 261 | 267 | 135 | 663
  UFH and/or LMWH: UFH | 221 | 236 | 120 | 577
  UFH and/or LMWH: LMWH | 25 | 24 | 10 | 59
  UFH and/or LMWH: UFH and LMWH | 15 | 7 | 5 | 27
  Another parenteral agent | 0 | 1 | 0 | 1
  None | 13 | 8 | 7 | 28
Time from study hospital presentation to treatment catheter insertion, hours [Mean (Standard Deviation); unit: hours] — Population: Data unavailable for 3 subjects in the Randomized Controlled Trial Cohort - FlowTriever Arm, 5 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm, and 3 subjects in the non-randomized cohort.
  hours
    number analyzed (Participants) | 271 | 271 | 139 | 681
    (all) | 22.3 (17.7) | 24.9 (19.7) | 38.3 (62.8) | 26.6 (33.4)
mPAP, mmHg [Mean (Standard Deviation); unit: mmHg] — Population: Data unavailable for 6 subjects in the Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm and 1 subject in the non-randomized cohort.
  mmHg
    number analyzed (Participants) | 274 | 270 | 141 | 685
    (all) | 30.0 (7.6) | 31.1 (7.2) | 29.7 (7.5) | 30.4 (7.4)

OUTCOME MEASURES:

1. Primary Outcome: Primary Endpoint: Composite Clinical Endpoint Constructed as a 5-Component Win Ratio
Description: The primary endpoint is a composite constructed as a hierarchical win ratio of the following 5 components:
  1. All-cause mortality, or
  2. Intracranial hemorrhage (ICH), or
  3. Major bleeding per ISTH definition, or
  4. Clinical deterioration defined by hemodynamic or respiratory worsening, and/or escalation to a bailout therapy, or
  5. ICU admission and ICU length-of-stay during the index hospitalization and following the index procedure.
  A win ratio larger than 1 indicates that patients who receive treatment with FlowTriever are more likely to have better outcomes as compared to subjects treated with CDT.
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: Enrolled subjects in the Randomized Controlled Trial Cohort - FlowTriever Arm and Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm were assessed for this Outcome Measure.
Measure: Number; unit: Number of Wins for the group
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm
Number analyzed (Participants) | 274 | 276
Number of Wins for the group | 52693 | 10509
Statistical Analysis 1: Comparison: Randomized Controlled Trial Cohort - FlowTriever Arm vs Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm; Test type: Superiority; Win Ratio = 5.01, 95% CI 2-sided [3.68 to 6.97]

2. Secondary Outcome: Composite Clinical Endpoint Constructed as a 4-Component Win Ratio
Description: This secondary endpoint is a composite constructed as a hierarchical win ratio of the following 4 components:
  * All-cause mortality, or
  * Intracranial hemorrhage (ICH), or
  * Major bleeding per ISTH definition, or
  * Clinical deterioration defined by hemodynamic or respiratory worsening, and/or escalation to a bailout therapy
  A win ratio larger than 1 indicates that patients who receive treatment with FlowTriever are more likely to have better outcomes as compared to subjects treated with CDT.
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: as for outcome 1
Measure: Number; unit: Number of Wins for the group
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm
Number analyzed (Participants) | 274 | 276
Number of Wins for the group | 7925 | 5912
Statistical Analysis 1: Comparison: Randomized Controlled Trial Cohort - FlowTriever Arm vs Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm; Test type: Superiority; Win Ratio = 1.34, 95% CI 2-sided [0.78 to 2.35]

3. Secondary Outcome: All-cause Mortality
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 276 | 142
Participants | 0 | 1 | 0

4. Secondary Outcome: Intracranial Hemorrhage (ICH)
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 275 | 142
Participants | 2 | 1 | 0

5. Secondary Outcome: Major Bleeding Per ISTH Definition
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 276 | 142
Participants | 19 | 19 | 10

6. Secondary Outcome: Clinical Deterioration Defined by Hemodynamic or Respiratory Worsening, and/or Escalation to a Bailout Therapy
Description: Clinical deterioration is defined as documented objective hemodynamic or respiratory worsening that is new (i.e. not present at the time of enrollment).
  Bailout therapy is an unplanned escalation of therapeutic measures, taken when the patient's condition has not improved or is not improving according to expectations.
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 276 | 142
Participants | 5 | 15 | 5

7. Secondary Outcome: ICU Admission During the Index Hospitalization and Following the Index Procedure
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 276 | 142
Participants | 114 | 272 | 65

8. Secondary Outcome: ICU Length of Stay During the Index Hospitalization and Following the Index Procedure Among Subjects With ICU Admission.
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 114 | 272 | 65
Participants
  ICU length of stay 0-24 hours | 61 | 94 | 30
  ICU length of stay >24 hours | 53 | 178 | 35

9. Secondary Outcome: All Cause Mortality
Time Frame: 30 days from index procedure
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 251 | 240 | 127
Participants | 1 | 2 | 5

10. Secondary Outcome: All-cause and PE-related Readmissions
Time Frame: 30 days from index procedure
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 251 | 239 | 124
Participants
  All-cause readmission | 8 | 19 | 13
  PE-related readmission | 0 | 2 | 1

11. Secondary Outcome: Device-related Serious Adverse Events
Description: Device-related SAEs included those adjudicated by the CEC to be related to the interventional device.
Time Frame: Through the 30 day visit
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 254 | 240 | 123
Participants | 19 | 12 | 9

12. Secondary Outcome: Drug-related Serious Adverse Events
Description: Drug-related SAEs included those adjudicated by the CEC to be related to anticoagulation and/or thrombolytics medication.
Time Frame: Through the 30 day visit
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 254 | 244 | 123
Participants | 31 | 28 | 18

13. Secondary Outcome: Clinically Relevant Non-Major (CRNM) and Minor Bleeding Events
Time Frame: Hospital discharge or at 7 days after the index procedure, whichever is sooner
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 275 | 142
Participants
  Clinically relevant non-major (CRNM) bleeding events | 7 | 9 | 6
  Minor bleeding events | 6 | 1 | 0

14. Secondary Outcome: Change in Right-ventricular/Left-ventricular (RV/LV) Ratio, as Measured by Echocardiography or CT
Description: Assessments of change were made using the same imaging modality at baseline and at the 24-hour visit.
Time Frame: Baseline to 24 hour visit
Population: All enrolled subjects with available outcome
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 259 | 259 | 127
ratio | -0.32 (0.24) | -0.30 (0.26) | -0.38 (0.29)

15. Secondary Outcome: Modified Medical Research Council (mMRC) Dyspnea Score at 24 Hour Visit
Description: The mMRC score is reported on a 0-4 scale with lower scores representing less dyspnea.
Time Frame: At 24 hour visit
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 259 | 250 | 130
Participants
  Score 0 - Dyspnea only with strenuous exercise | 80 | 77 | 40
  Score 1 - Dyspnea when hurrying or walking up a slight hill | 83 | 54 | 35
  Score 2 - Walks slower than people of the same age due to dyspnea or stops for breath when walking | 61 | 53 | 29
  Score 3 - Stops for breath after walking 100 yards (91 m) or after a few minutes | 27 | 44 | 21
  Score 4 - Too dyspneic to leave house or breathless when dressing | 8 | 22 | 5

16. Secondary Outcome: Modified Medical Research Council (mMRC) Dyspnea Score at 30 Day Visit
Description: The mMRC score is reported on a 0-4 scale with lower scores representing less dyspnea.
Time Frame: At 30 day visit
Population: All enrolled subjects with available outcome
Measure: Count of Participants; unit: Participants
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 258 | 254 | 121
Participants
  Score 0 - Dyspnea only with strenuous exercise | 137 | 138 | 60
  Score 1 - Dyspnea when hurrying or walking up a slight hill | 74 | 63 | 33
  Score 2 - Walks slower than people of the same age due to dyspnea or stops for breath when walking | 28 | 27 | 17
  Score 3 - Stops for breath after walking 100 yards (91 m) or after a few minutes | 14 | 23 | 6
  Score 4 - Too dyspneic to leave house or breathless when dressing | 5 | 3 | 5

17. Secondary Outcome: Length of Total Hospital Stay
Time Frame: Through 30 days post-procedure
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: hospital overnights
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 276 | 142
hospital overnights | 4.5 (2.8) | 5.3 (3.9) | 7.8 (7.4)

18. Secondary Outcome: Length of Post-index-procedure Hospital Stay
Time Frame: Through 30 days post-procedure
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 274 | 276 | 142
days | 3.2 (2.72) | 4.0 (3.71) | 5.4 (5.80)

19. Secondary Outcome: Pulmonary Embolism Quality of Life (PEmb-QOL) Score at 30 Day Visit
Description: The Pulmonary Embolism Quality of Life (PEmb-QOL) questionnaire is used to assess the quality of life in patients with pulmonary embolism (PE). It is a disease-specific tool designed to evaluate the impact of PE on various aspects of a patient's life, including daily activities, work, social life, and emotional well-being, and is reported on a 0-100 scale with lower scores representing better quality of life.
Time Frame: At 30 day visit
Population: All enrolled subjects with available outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 260 | 253 | 123
score on a scale | 19.33 (18.91) | 20.42 (19.95) | 23.50 (21.75)

20. Secondary Outcome: EQ-5D-5L Quality of Life Score at 30 Day Visit
Description: Each of the five dimensions comprising the EQ-5D-5L descriptive system (mobility, self-care, usual activates, pain/discomfort, anxiety/depression) are graded from 1 (no problems) to 5 (extreme problems). A descriptive health state is defined by combining each level for 5 dimensions into a 5-digit code (e.g., 12345) which is then mapped to the health state index score based on a country-specific value set. Health state index scores range from less than 0 (where 0 is the value of a health state equivalent to dead; negative values representing values as worse than dead) to 1 (the value of full health).
Time Frame: At 30 day visit
Population: All enrolled subjects with available outcome
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
Number analyzed (Participants) | 259 | 255 | 123
score on a scale | 0.829 (0.218) | 0.817 (0.237) | 0.742 (0.284)

ADVERSE EVENTS:
Time Frame: Adverse events collected from time of enrollment through 30 Day visit or study exit, if exited early. For European subjects, reporting began after signing informed consent, while US subjects reporting began after the study device entered the vasculature. The All-Cause Mortality field reports all deaths reported through study exit and from vital status tracing after exit (including cases of sponsor awareness after exit), differing slightly from the 30-day all-cause mortality secondary endpoint.
Description: All CEC adjudicated events (all SAEs and non-serious AEs potentially related to a primary/secondary endpoint reported prior to study exit) as well as non-adjudicated events known from vital status tracing in subjects lost to follow-up are listed here. Mortality status is known at the earlier of study exit or day 30 for everyone except 2 RCT subjects lost to follow-up. The all-cause mortality rate excluding these subjects is 1.1% (3/273) for the FlowTriever arm and 0.7% (2/275) for the CDT arm.
Arm/Group | Randomized Controlled Trial Cohort - FlowTriever Arm | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm | Non-Randomized Absolute Contraindication to Thrombolytics Cohort
All-Cause Mortality (participants affected / at risk) | 3/274 | 2/276 | 6/142
Serious Adverse Events (participants affected / at risk) | 43/274 | 47/276 | 35/142
Other Adverse Events (participants affected / at risk) | 23/274 | 18/276 | 13/142
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Controlled Trial Cohort - FlowTriever Arm (N=274) | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm (N=276) | Non-Randomized Absolute Contraindication to Thrombolytics Cohort (N=142)
Deep vein thrombosis (Vascular disorders) | 2 | 1 | 1
Hypotension (Vascular disorders) | 2 | 3 | 1
Syncope (Vascular disorders) | 2 | 0 | 0
Abdominal wall haematoma (Vascular disorders) | 1 | 0 | 0
Cerebral haemorrhage (Vascular disorders) | 1 | 1 | 0
Cerebrovascular accident (Vascular disorders) | 1 | 0 | 2
Haematoma (Vascular disorders) | 1 | 0 | 0
Heparin-induced thrombocytopenia (Vascular disorders) | 1 | 0 | 1
Postmenopausal haemorrhage (Vascular disorders) | 1 | 0 | 0
Pulmonary embolism (Vascular disorders) | 1 | 4 | 1
Chest wall haematoma (Vascular disorders) | 0 | 1 | 0
Embolic stroke (Vascular disorders) | 0 | 0 | 1
Gangrene (Vascular disorders) | 0 | 0 | 1
Haematoma muscle (Vascular disorders) | 0 | 1 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 0 | 1
Iliac artery occlusion (Vascular disorders) | 0 | 1 | 0
Presyncope (Vascular disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 0 | 1 | 0
Thrombosis (Vascular disorders) | 0 | 0 | 1
Vascular access site haematoma (Injury, poisoning and procedural complications) | 7 | 7 | 1
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 3 | 1 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0 | 0
Catheter site haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 1
Orbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative wound infection (Injury, poisoning and procedural complications) | 0 | 0 | 1
Procedural hypotension (Injury, poisoning and procedural complications) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 5
Blood loss anaemia (Blood and lymphatic system disorders) | 1 | 1 | 3
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Normocytic anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Dyspnoea (Cardiac disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 0 | 0 | 2
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Intra-abdominal haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Mesenteric neoplasm (Gastrointestinal disorders) | 0 | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 1
Septic shock (Infections and infestations) | 1 | 1 | 2
Pneumonia (Infections and infestations) | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 3 | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1 | 0
Renal transplant failure (Renal and urinary disorders) | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 2 | 2 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Alcohol withdrawal syndrome (General disorders) | 0 | 1 | 0
Chest pain (General disorders) | 0 | 2 | 0
Death (General disorders) | 0 | 1 | 0
Generalised oedema (General disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0
Vessel puncture site haematoma (General disorders) | 0 | 2 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0 | 0
Biliary dilatation (Hepatobiliary disorders) | 0 | 0 | 1
Toxic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 2 | 0
Catheter directed thrombolysis (Surgical and medical procedures) | 1 | 0 | 0
Thrombectomy (Surgical and medical procedures) | 1 | 1 | 0
Arterial puncture (Surgical and medical procedures) | 0 | 0 | 1
Lung assist device therapy (Surgical and medical procedures) | 0 | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteorrhagia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Randomized Controlled Trial Cohort - FlowTriever Arm (N=274) | Randomized Controlled Trial Cohort - Catheter-Directed Thrombolysis Arm (N=276) | Non-Randomized Absolute Contraindication to Thrombolytics Cohort (N=142)
Vascular access site haemorrhage (Injury, poisoning and procedural complications) | 6 | 0 | 0
Vascular access site haematoma (Injury, poisoning and procedural complications) | 3 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Non-small cell lung cancer (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Bradycardia (Cardiac disorders) | 1 | 0 | 1
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 1
Pericardial effusion (Cardiac disorders) | 0 | 2 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 1 | 0 | 0
Pharyngo-oesophageal diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
Cerebrovascular accident (Vascular disorders) | 0 | 0 | 1
Epistaxis (Vascular disorders) | 0 | 1 | 0
Swelling face (General disorders) | 1 | 0 | 0
Necrosis (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 1 | 0
Right ventricular systolic pressure decreased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 1 | 0
Oxygen saturation decreased (Investigations) | 0 | 1 | 0
Respiratory rate increased (Investigations) | 0 | 1 | 0
Transaminases increased (Investigations) | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 2 | 0
Blood loss anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Metastatic uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Abortion induced (Surgical and medical procedures) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2023-08-23): https://cdn.clinicaltrials.gov/large-docs/13/NCT05111613/Prot_000.pdf
  • Statistical Analysis Plan (2024-03-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT05111613/SAP_001.pdf